CLINICAL TRIAL: NCT06667609
Title: Validity and Reliability of the Mastitis Symptom Severity Assessment Methods (M-Score and BISSI) in Non-Lactational Mastitis
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Chen Kai, Vice Director of Dept Breast Surgery., Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSKY-2024-699-01
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Granulomatous Mastitis; Mastitis Chronic
Keywords: M-score; validity; reliability
MeSH Terms: conditions — Granulomatous Mastitis | interventions — Surgical Procedures, Operative; Adrenal Cortex Hormones; Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 1: This is an observational study with no predefined treatments for the enrolled patients. Participants may receive any treatments in accordance with standard clinical practice, based on physicians' recommendations and patients' preferences.
  Interventions: Other: Any treatments regimen

INTERVENTIONS:
Other: Any treatments regimen — Participants may receive any treatments in accordance with standard clinical practice, based on physicians' recommendations and patients' preferences.
  Other Names: Surgery; Corticosteroids; Ductal lavage; Anti-TB treatments; Observations; Aspirations; Immuno-suppression medications

SUMMARY:
The purpose of this study is to evaluate the validity and reliability of the Mastitis-score (M-score) and the Breast Inflammatory Symptom Severity Index (BISSI) as measures for assessing symptom severity in non-lactational granulomatous lobular/periductal mastitis (NL-GLM/PDM). This research aims to provide a valid and reliable tool for evaluating both symptom severity and treatment efficacy in NL-GLM/PDM.

DETAILED DESCRIPTION:
Non-lactational granulomatous lobular/periductal mastitis (NL-GLM/PDM) are inflammatory breast diseases with unclear etiology, usually manifested as palpable breast mass, accompanied by breast pain and abscesses, erythema or fistula formation. There is no well-recognized assessment tool for evaluating the symptom severity and treatment efficacy of NL-GLM/PDM. In our previous studies with NL-GLM, we used the Mastitis-score (M-score) as a physician-directed measure of the symptom severity. However, there were no patient-reported outcome measure for NL-GLM/PDM. The Breast Inflammatory Symptom Severity Index(BISSI) was reported as a valid patient-reported outcome measure for lactational mastitis. Its clinical validity as a measure of Symptom Severity for NL-GLM/PDM are still unclear.

In this multicenter, prospective cohort study, we will validate the validity and reliability of the M-score, a physician-directed measure, and the Breast Inflammatory Symptom Severity Index (BISSI), a patient-reported outcome (PRO) measure, for assessing symptom severity in patients with non-lactational granulomatous lobular/periductal mastitis (NL-GLM/PDM). Establishing the validity of these two approaches will facilitate the objective measurement of treatment efficacy for NL-GLM/PDM in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Female, age between 18 and 65 years;
2. Clinically considered as Non-Lactational mastitis;
3. Clinically and Pathologically confirmed NL-GLM/PDM;
4. Patients planning to receive treatment or observation alone;
5. Signed the informed consent form

Exclusion Criteria:

1. Patients with confirmed or suspected malignant breast tumors
2. Patients with bilateral mastitis (including those with bilateral Non-Lactational Mastitis occurring simultaneously or successively)
3. Pregnant.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female diagnosed with NL-GLM/PDM in China
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Inter-rater Reliability | 8 weeks
  This assesses the consistency of results from different evaluators regarding the various dimensions of the Mscore and the total M-score for the same patients at the same time.
Test-Retest Reliability | 8 weeks
  This assesses the consistency of the M-score/BISSI results for the same patient at different times (within 1 week after enrollment), prior to treatment initiation and when symptoms have not changed significantly.
Clinical Validity | 8 weeks
  This aims to estimate the correlation between the M-score/BISSI and its changes, and the BISSI and its changes, with traditional evaluator assessments or traditional patient self-assessments of treatment efficacy and its changes.

SECONDARY OUTCOMES:
Correlation between the M-score/BISSI with laboratory indicators | 8 weeks
  Explore the correlation between the M-score/BISSI with white blood cell counts, neutrophil counts, lymphocyte counts, neutrophil/lympocyte ratio, CRP, ESR, TNF-alpha, and IL-6.
Cutoff value for M-score/BISSI to defined clinical complete remission. | 8 weeks
  Investigate the optimal cutoff value of the M-score/BISSI for defining clinical complete remission.
Correlation between the M-score and BISSI scores. | 8 weeks
  Examine the correlation between the M-score and BISSI scores.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Chaozhou Maternal and Child Health Hospital, Chaozhou, Guangdong
  - Dongguan Maternal and Child Health Care Hospital, Dongguan, Guangdong
  - Sun Yat-sen memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Jiangmen Maternity and Child Health Care Hospital, Jiangmen, Guangdong
  - Shenshan Medical Center, Sun Yat-sen Memorial Hospital, Shanwei, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided
If the study can be completed and the data have been collected, sharing IPD with the approval from the administrator would be feasible.

REFERENCES:
- [Background] Heron E, McArdle A, Karim MN, Cooper M, Geddes D, McKenna L. Construct validity and internal consistency of the Breast Inflammatory Symptom Severity Index in lactating mothers with inflammatory breast conditions. PeerJ. 2021 Nov 16;9:e12439. doi: 10.7717/peerj.12439. eCollection 2021. PMID 34820185
- [Background] Chen X, Huang H, Huang H, Yong J, Zhu L, Chen Q, Tan L, Zeng Y, Yang Y, Zhao J, Rao N, Ding L, Wu W, Li Y, Gui X, Ye L, Xu Y, Jiang Y, Su L, Xiao Q, Cai X, Hu T, Tan C, Liu Q, Liu S, Zhao J, Wang Y, Yu F, Zhang J, Li S, Chen K. Ductal lavage followed by observation versus oral corticosteroids in idiopathic granulomatous mastitis: A randomized trial. Nat Commun. 2024 Oct 23;15(1):9144. doi: 10.1038/s41467-024-53143-2. PMID 39443446